CLINICAL TRIAL: NCT04657549
Title: Partial or Total Surgical Removal of Palatal Tonsils to Change Quality of Life for Adults With Chronic or Recurrent Tonsillitis: Randomized Controlled Trial.
Brief Title: Tonsil Surgery in Recurrent or Chronic Tonsillitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Olli-Pekka Alho, MD, Professor, MD, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Diary number 113/2020
Record Dates: First submitted 2020-11-16; First posted 2020-12-08 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Tonsillitis Recurrent; Tonsillitis Chronic
Keywords: tonsillitis; tonsillectomy; tonsillotomy; tonsil surgery
MeSH Terms: conditions — Tonsillitis | interventions — Tonsillectomy; sipuleucel-T

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients in active arms don't know if they are in tonsillectomy or tonsillotomy group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tonsillectomy (Active Comparator): Patients will undergo tonsillectomy under general anesthesia within three weeks after enrollment.
  Interventions: Procedure: Tonsillectomy
- Tonsillotomy (Active Comparator): Patients will undergo tonsillotomy under general anesthesia within three weeks after enrollment.
  Interventions: Procedure: Tonsillotomy
- Watchful waiting (No Intervention): Patients will be closely monitored for the 5-6 months monitoring period.

INTERVENTIONS:
Procedure: Tonsillectomy — Tonsillectomy is done by monopolar electrocautery, bipolar scissors or cold instruments. First the mucosa of the anterior palatinal arch is incised and tonsillar capsule identified, then tonsillar tissue is removed along the capsule. Any bleeding is coagulated either with monopolar or bipolar electrocautery.
  Other Names: Extracapsular tonsillectomy, ECTE
  Arms: Tonsillectomy
Procedure: Tonsillotomy — Tonsillotomy is done using monopolar electrosurgery, bipolar scissors or coblator device. Most of the tonsillar tissue is removed, exceeding the removal behind the line between anterior and posterior palatinal arch so that only thin layer of tonsil tissue is left over the tonsillar capsule.
  Other Names: Intracapsular tonsillectomy, ICTE. Subtotal/intracapsular/partial tonsillectomy, SIPT.
  Arms: Tonsillotomy

SUMMARY:
Tonsil surgery is common in adults with recurrent or chronic tonsillitis. The surgical techniques include either partial or total surgical removal of the palatal tonsils (tonsillotomy, TT, and tonsillectomy, TE, respectively). The aim of this study is to find out, whether tonsil surgery improves the quality of life in these patients and whether the lighter TT is as effective as TE. Our main outcome is the disease-specific Tonsillectomy Outcome Inventory-14 (TOI-14) quality of life questionnaire score at 6 months follow-up.

DETAILED DESCRIPTION:
Rationale

Surgical removal of palatal tonsils is among the most common ear, nose and throat operations in adults in Finland. The vast majority of these operations are done for recurrent and chronic tonsillitis. Internationally accepted guidelines for the treatment of these diseases are lacking and the indications for tonsil surgery are practice-based rather than evidence-based. The choice of the surgical technique further confuses the picture. The traditional surgical technique has been the total removal of tonsils (tonsillectomy, TE). The relatively recent introduction of partial resection of tonsils, namely tonsillotomy (TT), is suggested to have the benefits of less postoperative pain and smaller risk of post-operative hemorrhage as compared to TE. The relative efficacy of these two techniques to alleviate infective tonsillar diseases is still unclear.

Objectives

The main aim of this study is to obtain reliable evidence on, whether tonsil surgery improves the quality of life in adult patients suffering from recurrent or chronic tonsillitis, and whether the lighter TT would be as effective as TE. We will also compare the scores of a generic quality of life questionnaire as well as several other subjective and objective beneficial and harmful outcomes between the groups.

Methods

In this pragmatic multi-center randomized controlled trial, adult patients suffering from recurrent or chronic tonsillitis will be randomly allocated to three groups: tonsillotomy group (TT), tonsillectomy group (TE) and control group with watchful waiting (WW) in ratio 2:2:1. The patients in the surgical groups are blinded to the operation type (TT or TE). Our hypothesis is that both surgical treatments are more effective than watchful waiting in enhancing quality of life without significant risks (superiority assumption) and that TT is non-inferior to TE when the surgical groups are compared (non-inferiority assumption). Our principal outcome is disease-specific quality of life questionnaire score (Tonsillectomy Outcome Inventory (TOI)-14) at 6 months follow-up. We have validated this questionnaire in Finnish and explored the interpretation of the scores. Secondary outcomes have been listed in the Outcomes section.

Separate random allocation lists for the main research center (Oulu University Hospital) and for the four other centers collectively as well as for recurrent and for chronic tonsillitis will be used. Random permuted blocks is used with block size varying between 5 and 10. Based on our earlier study, the principal outcome, TOI-14 score, will most probably be left-truncated at zero and right-skewed. Therefore, both tobit-analysis and covariate analysis is used with log (1+y) transformation. The primary analysis has two phases. Firstly, the TOI-14 score in the combined surgical group (TT+TE) is compared to that in the WW group. Secondly, the score in the TT group is compared to that in the TE group. Effects will be estimated by adjusted mean differences in the log-transformed scores with 95% confidence intervals. Based on our earlier observational studies on the subject, the following covariates are included in the multivariable adjusted model: gender and baseline TOI-14 score together with stratification factors: enrolling center (Oulu vs. others) and main complaint (recurrent vs. chronic tonsillitis). In case there is missing data on the primary outcome, a multiple imputation method will be used. The analyses will be performed on an intention to treat basis. Per protocol analysis will be performed as sensitivity analysis and results from comparisons on secondary outcomes and subgroup analysis (main complaint) are used to generate hypothesis for future trials.

ELIGIBILITY:
The inclusion criteria are:

* Recurrent tonsillitis episodes:

  * At least 4 episodes in the previous 12 months or at least 3 episodes in 6 months
  * Episodes are disabling, prevent normal functioning and are severe enough for the patient to seek medical attention
  * Episodes are thought to involve the palatine tonsils based on signs found during the episodes (e.g. edema, erythema, exudative tonsillitis, anterior cervical lymphadenitis)
  * No throat cultures or antigen/molecular tests to show infection with group A streptococcus are needed
* Chronic tonsillitis:

  * Recurrent or chronic throat pain for at least 6 months
  * At least one symptom or sign that indicate that symptoms originate from the palatal tonsils (disturbing tonsil stones, halitosis, anterior cervical lymphadenitis, tonsillar exudates, abnormal tonsillar crypts)
  * Symptomatic treatment has not been effective

The exclusion criteria are:

* Age less than 18 years
* Pregnancy
* History of peritonsillar abscess
* Previous illness that make prompt same-day surgery unfeasible
* No electronic identity verification tools

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Tonsillectomy Outcome Inventory -14 (TOI-14) follow-up score | At the end of five to six months follow-up
  TOI-14 is a disease-specific quality of life questionnaire for throat related symptoms in adults. TOI-14 summary scores vary between 0 and 100 with higher values indicating poorer quality of life. Analysis is described in the Detailed Description section.

SECONDARY OUTCOMES:
36-Item short Form Survey (SF-36, RAND-36) follow-up score | At the end of five to six months follow-up
  Difference in RAND-36 domains scores between groups. RAND-36 instrument produces eight individual values between 0 and 100 (one for each domain), with higher scores indicating better quality of life
Proportion benefiting | At the end of five to six months follow-up
  Difference in proportions of patients benefiting clinically significantly from the intervention between the groups (minimum important change in TOI-14 score)
Days with throat pain | At the end of five to six months follow-up
  Difference in the number of days patients have throat pain (severity scaled 0-10) between the groups
Days with halitosis | At the end of five to six months follow-up
  Difference in the number of days patients have bad breath (severity scaled 0-10) between the groups
Days with bleeding | At the end of five to six months follow-up
  Difference in the number of days patients have bleeding from the throat (severity scaled 0-10) between the groups
Days with tonsil stones | At the end of five to six months follow-up
  Difference in the number of days patients have bothering tonsil stones (severity scaled 0-10) between the groups
Days with absence from work | At the end of five to six months follow-up
  Difference in the number of days patients are absent from work or school due to throat symptoms between the groups
Days with dexketoprofen | At the end of five to six months follow-up
  Difference in the number of days patients take deksketoprofen 25 mg pain medication due to throat pain between the groups
Days with acetaminophen | At the end of five to six months follow-up
  Difference in the number of days patients take acetaminophen 1 g pain medication due to throat pain between the groups
Days with oxycodone/naloxone | At the end of five to six months follow-up
  Difference in the number of days patients take oxycodone/naloxone 5mg/2.5mg pain medication due to throat pain between the groups
Medical visits | At the end of five to six months follow-up
  Difference in the number of medical visit for throat symptoms between the groups
Antibiotic courses | At the end of five to six months follow-up
  Difference in the number of antibiotic courses for throat symptoms between the groups
Adverse effect-postoperative bleeding | At the end of five to six months follow-up
  Frequency of postoperative bleeding in the surgical groups
Adverse effect - postoperative pain | At the end of five to six months follow-up
  Frequency of postoperative pain in the surgical groups
Adverse effect - postoperative infection | At the end of five to six months follow-up
  Frequency of postoperative infections in the surgical groups
Adverse effect - dental injury | At the end of five to six months follow-up
  Frequency of dental injury in the surgical groups
Adverse effect -anesthetic complication | At the end of five to six months follow-up
  Frequency of anesthetic complication in the surgical groups
Adverse effect - tightness/globus | At the end of five to six months follow-up
  Difference in proportions having feeling of tightness/globus in throat between the groups
Adverse effect - voice problems | At the end of five to six months follow-up
  Difference in proportions having voice problems between the groups
Adverse effect - jaw problems | At the end of five to six months follow-up
  Difference in proportions having mandibular joint problems between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Olli-Pekka Alho, MD, PhD, Principal Investigator — Oulu University Hospital, University of Oulu; Aleksi EJ Laajala, MD, Study Chair — Oulu University Hospital, University of Oulu; Paulus Tokola, MD, Study Chair — Oulu University Hospital, University of Oulu; Timo J Autio, MD, PhD, Study Chair — Oulu University Hospital; Timo J Koskenkorva, MD, PhD, Study Chair — University of Oulu; Pasi Ohtonen, M. Sc., Study Chair — Division of Operative Care, Oulu University Hospital, Finland; Esa Läärä, PhD., Study Chair — Oulu University
Locations (7):
- Finland (7):
  - Lapland Central Hospital, Rovaniemi, Lapland
  - Länsi-Pohja Central Hospital, Kemi
  - Keski-Pohjanmaa Central Hospital, Kokkola
  - Oulu University Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki
  - Turun yliopistollinen keskussairaala, Turku
  - Vaasan keskussairaala, Vaasa

IPD SHARING:
Plan to Share IPD: Yes
Study protocol that includes the Informed Consent Form will be sent to a journal for publication, Statistical analysis Plan will be published later in ClinicalTrials.gov web site.
  The data generated or analyzed during this study will be available from the corresponding investigator on reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol will be sent for publication within 12 months from the beginning of recruiting. Data from the study will be available starting six months after publication.
Access Criteria: The data generated or analyzed during this study will be available from the corresponding investigator on reasonable request.

REFERENCES:
- [Background] Laajala A, Autio TJ, Ohtonen P, Alho OP, Koskenkorva TJ. Interpretation of Tonsillectomy Outcome Inventory-14 scores: a prospective matched cohort study. Eur Arch Otorhinolaryngol. 2020 May;277(5):1499-1505. doi: 10.1007/s00405-020-05832-z. Epub 2020 Feb 14. PMID 32060601
- [Background] Koskenkorva T, Koivunen P, Laara E, Alho OP. Predictive factors for quality of life after tonsillectomy among adults with recurrent pharyngitis: a prospective cohort study. Clin Otolaryngol. 2014 Aug;39(4):216-23. doi: 10.1111/coa.12263. PMID 24863677
- [Background] Laajala A, Tokola P, Autio TJ, Koskenkorva T, Tastula M, Ohtonen P, Laara E, Alho OP. Total or partial tonsillar resection (tonsillectomy or tonsillotomy) to change the quality of life for adults with recurrent or chronic tonsillitis: study protocol for a randomised controlled trial. Trials. 2021 Sep 15;22(1):617. doi: 10.1186/s13063-021-05539-4. PMID 34526073

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT04657549/SAP_000.pdf